CLINICAL TRIAL: NCT05385354
Title: Normal Values of Main Pancreatic Duct Diameter
Brief Title: Main Pancreatic Duct Diameter
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Veit Phillip, Senior physician, head of clinical pancreatology, Technical University of Munich
Other Study IDs: MDP-1
Record Dates: First submitted 2022-05-06; First posted 2022-05-23 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Duct Dilatation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The maximal diameter of the pancreatic duct will be measured by endoscopic ultrasound at four different parts:

* Pancreatic head
* Pancreatic neck
* Pancreatic body
* Pancreatic tail

DETAILED DESCRIPTION:
All patients without pancreatic or biliary disorders undergoing upper-GI endoscopic ultrasound (EUS) are eligible for the study.

The maximal diameter of the pancreatic duct will be measured by endoscopic ultrasound in millimeters at four different parts:

* Pancreatic head
* Pancreatic neck
* Pancreatic body
* Pancreatic tail

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing EUS for investigation of non-pancratic disease (e.g. subeptithelial tumor of the upper GI-tract
* Indication for EUS is undependent from the study
* Written informed consent
* Age ≥18 years

Exclusion Criteria:

* Pancreatic diseases (chronic or acute pancreatitis, pancreatic tumor, pancreatic cyst, etc.)
* Disorders of papilla duodeni major/minor (adenoma/carcinoma of papilla duodeni major or minor)
* Biliary disorders (bile duct stones, cholangio carcinoma, cholangitis)
* Elevated Bilirubin and/or Lipase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing EUS for investigation of non-pancratic disease (e.g. subeptithelial tumor of the upper GI-tract
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Maximal diameter of main pancreatic duct in millimeters | The measurement is performed once during endosonography.
  Measurements of main pancreatic duct at different sections of the pancreas

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic and Policlinik of Internal Medicine II, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided